CLINICAL TRIAL: NCT01773135
Title: Maternal Serum Level of ACTH as a Predictive Marker of Preterm Labor in Patients With Threatened Preterm Labor
Acronym: PTL
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Saied Eldein El-Safty, Lecturer of Obstetrics and Gynecology Faculty of Medicine - Ain Shams University, Ain Shams Maternity Hospital
Other Study IDs: mai-01110333535; MAI-01110333535m (Registry Identifier: mai ibrahim ali ibrahim)
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Threatened Preterm Labor
Keywords: threatened preterm labor; ACTH; PTL

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Weeks
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- preterm group: pregnant healthy women aged from 17 to 35 who suffered from symptoms of threatened preterm labor in the form of Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes), Cervical dilation > 1 and < 4 cm, and/or Cervical effacement ≥ 80%. collection of blood sample and tocolysis administration will be done this group will deliver preterm (before 37 weeks of gestation)
  Interventions: Other: collection of blood sample and tocolysis adminstration
- full term group: pregnant healthy women aged from 17 to 35 who suffered from symptoms of threatened preterm labor in the form of Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes), Cervical dilation > 1 and < 4 cm, and/or Cervical effacement ≥ 80%. collection of blood sample and tocolysis administration will be done this group will deliver full term (after 37 weeks of gestation)
  Interventions: Other: collection of blood sample and tocolysis adminstration

INTERVENTIONS:
Other: collection of blood sample and tocolysis adminstration — investigators will abtain a blood sample from all patient to measure the serum level of ACTH.
  all patients with threatened preterm labor will receive a fixed regimen of tocolysis in the form of nifedipine (Epilate) 10 mg orally every 15 minutes for the first hour or until cessation of uterine contractions. Then, 60 - 160 mg/day (1-2 tablets 3 times daily) of slowly releasing nifedipine (epilat retard 20 mg tablet) may be given depending on uterine activity. The patients will also receive 6 mg dexamethasone every 12 hours for 4 doses. All women will be followed up till delivery.
  After delivery, investigators devide the pateints into 2 groups (full term delivery & preterm delivery) and investigators compare between these 2 groups by level of hormone.

SUMMARY:
The aim of this study is use of ACTH as a predictive marker in patients of threatened preterm labor .

DETAILED DESCRIPTION:
This is a cross sectional study that will include 261 pregnant women aged between 17 and 35 years with singleton pregnancies between 28 and 36 completed weeks of gestation that had been diagnosed with threatened preterm labor and consented to participate in this study. This study will be conducted at Ain Shams University Maternity Hospital after approval of the research and ethics committee.

the investigators include all patients which have these following criteria (Singleton pregnancy, Age between 17 - 35 years, Gestational age between 28 and 36 weeks and Diagnosis of threatened preterm labor is based on the American College of Obstetricians and Gynaecologists Guidelines (ACOG, 2003): Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes), Cervical dilation > 1 and < 4 cm, and/or Cervical effacement ≥ 80%.

the investigators exclude any patient which has any of the following criteria (Preterm rupture of membranes, Any uterine anomalies or cervical incompetence, Chronic illness such as chronic hypertension or kidney disease, Diabetes mellitus, Abruptio placenta, Preeclampsia and HELLP syndrome, Fetal anomalies, IUGR, Smoking or Clinical signs of intrauterine infection).

blood sample was collected from each patient for measurement of ACTH level. According to local protocol in Ain Shams University Maternity Hospital all women will receive a fixed regimen of tocolysis in the form of nifedipine (Epilat) 10 mg orally every 15 minutes for the first hour or until cessation of uterine contractions. Then, 60 - 160 mg/day (1-2 tablets 3 times daily) of slowly releasing nifedipine (epilat retard 20 mg tablet) may be given depending on uterine activity. The patients will also receive 6 mg dexamethasone every 12 hours for 4 doses. All women will be followed up till delivery.

After delivery, the investigators divide the patients into 2 groups (full term delivery & preterm delivery) and we compare between these 2 groups by level of hormone.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Age between 17 - 35 years.
* Gestational age between 28 and 36 weeks.
* Diagnosis of threatened preterm labor is based on the American College of Obstetricians and Gynaecologists Guidelines (ACOG, 2003): Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes), Cervical dilation > 1 and < 4 cm, and/or Cervical effacement ≥ 80%.

Exclusion Criteria:

* Preterm rupture of membranes.
* Any uterine anomalies or cervical incompetence.
* Chronic illness such as chronic hypertension or kidney disease.
* Diabetes mellitus.
* Abruptio placenta.
* Preeclampsia and HELLP syndrome.
* Fetal anomalies.
* IUGR.
* Smoking.
* Clinical signs of intrauterine infection eg (uterine tenderness, foul vaginal discharge, maternal pyrexia ≥ 38°C and/or maternal leucocytosis).

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant women aged between 17 and 35 years with singleton pregnancies between 28 and 36 completed weeks of gestation that had been diagnosed with threatened preterm labor
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Elsafty, M.D., Principal Investigator — Ain Shams University
Locations (1):
- Ainshams Maternity hospital, Cairo, Egypt, Egypt

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women With Threatened Preterm Labor: pregnant healthy women aged from 17 to 35 who suffered from symptoms of threatened PTL in the form of Presence of uterine contractions (at least 4 in 20 minutes or 8 in 60 minutes), Cervical dilation > 1 and < 4 cm, and/or Cervical effacement ≥ 80%.
  then, collection of blood sample and tocolysis adminstration will be done
  investigators obtained a blood sample from all patient to measure the serum level of ACTH.
  all patients with threatened preterm labor will received a fixed regimen of tocolysis in the form of nifedipine (Epilate) 10 mg orally every 15 minutes for the first hour or until cessation of uterine contractions. Then, 1-2 tablets 4 times daily of slowly releasing nifedipine (epilat retard 20 mg tablet). All women will be followed up till delivery.
  After delivery, investigators devide the pateints into 2 groups (full term delivery & preterm delivery) and investigators compare between these 2 groups by level of hormone.
Period: Overall Study
Arm/Group | Pregnant Women With Threatened Preterm Labor
Started | 262
Completed | 262
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Preterm Group: pregnant healthy female aged from 17 to 35 who suffered from symptoms of threatened preterm labor.
  investigators obtained a blood sample from all patient to measure the serum level of ACTH.
  all patients with threatened preterm labor received a fixed regimen of tocolysis in the form of nifedipine (Epilate) 10 mg orally every 15 minutes for the first hour or until cessation of uterine contractions. Then, 60 - 160 mg/day (1-2 tablets 3 times daily) of slowly releasing nifedipine (epilat retard 20 mg tablet). The patients will also receive 6 mg dexamethasone every 12 hours for 4 doses. All women followed up till delivery.
  this group delivered preterm (before 37 weeks of gestation)
- Full Term Group: pregnant healthy female aged from 17 to 35 who suffered from symptoms of threatened preterm labor.
  investigators obtained a blood sample from all patient to measure the serum level of ACTH.
  all patients with threatened preterm labor received a fixed regimen of tocolysis in the form of nifedipine (Epilate) 10 mg orally every 15 minutes for the first hour or until cessation of uterine contractions. Then, 60 - 160 mg/day (1-2 tablets 3 times daily) of slowly releasing nifedipine (epilat retard 20 mg tablet). The patients will also receive 6 mg dexamethasone every 12 hours for 4 doses. All women followed up till delivery.
  this group delivered full term (after 37 weeks of gestation)
- Total: Total of all reporting groups
Arm/Group | Preterm Group | Full Term Group | Total
Number analyzed (Participants) | 161 | 101 | 262
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 29] | 26 [22 to 30] | 26 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 101 | 262
  Male | 0 | 0 | 0
gestational age at admission [Median (Inter-Quartile Range); unit: weeks] | 31 [29 to 33] | 31 [30 to 33] | 31 [30 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Evaluate if ACTH Can be Used as a Predictive Marker for Preterm Labor
Description: measurement of maternal serum ACTH in women daignosed as threatened preterm labor to evaluate if this hormone can be used as a predictive marker for preterm labor
Time Frame: 9 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Preterm Group: group of patients who delivered before 37 weeks of gestation
- Full Term Group: group of patients who delivered after 37 weeks of gestation
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 161 | 101
pg/ml | 23.4 [19.2 to 29] | 19.3 [16.7 to 21.5]
Statistical Analysis 1: Comparison: Preterm Group vs Full Term Group; Test type: Superiority or Other; p < 0.001, U statistic

ADVERSE EVENTS:
Arm/Group | Pregnant Women With Threatened Preterm Labor
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
It's the different time of day that blood sampling was carried out, although this reflects normal clinical practice, blood samples were collected at the time of admission to hospital regardless of the time of day, rather than diurnal pattern of ACTH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes